CLINICAL TRIAL: NCT00206869
Title: Does Exercise and Heat Increase the Lightsensibility in Patients With Erythropoietic Protoporphyria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KF 01-169/02
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2002-12

CONDITIONS: Erythropoietic Protoporphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — Exercise; Hot Temperature

INTERVENTIONS:
Behavioral: exercise
Behavioral: heat
Procedure: red light illumination

SUMMARY:
The purpose of the study is to evaluate the effect of exercise and heat on the light sensibility of patients with erythropoietic protoporphyria

ELIGIBILITY:
Inclusion Criteria: erythropoietic protoporphyria, age 14 to 70.

-

Exclusion Criteria:

* Not able to exercise

Ages: 14 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Wulf, MD, Sci, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark